CLINICAL TRIAL: NCT01817309
Title: Bacteria Endotoxin in Peritoneal Dialysis Effluent as a Predictor of Relapsing, Recurrent, and Repeat Peritonitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BLPS
Record Dates: First submitted 2013-03-19; First posted 2013-03-25 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Peritoneal Dialysis Associated Peritonitis
Keywords: renal failure; survival; peritoneal failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): endotoxin assay in peritoneal dialysis effluent
  Interventions: Other: endotoxin assay in peritoneal dialysis effluent

INTERVENTIONS:
Other: endotoxin assay in peritoneal dialysis effluent — endotoxin level by Limulus Amebocyte Lysate (LAL) assay

SUMMARY:
Peritoneal dialysis (PD) is the first-line treatment of end stage renal disease (ESRD) in Hong Kong. Despite the advances in antibiotic therapy and connecting system, recurrent peritonitis remains the major cause of peritoneal failure. A reliable predictor of relapsing peritonitis is invaluable in the management of PD peritonitis. Recent studies showed that bacterial-derived lipopolysaccharide (LPS) fragments are present in clinically used fluids such as dialysis fluid. LPS are thought to be derived from microorganisms inhabiting body fluid. The investigators hypothesize that the presence of LPS in PD effluent is a predictor of relapsing peritonitis in PD patients. The investigators plan to study 300 patients with PD peritonitis. After inform consent, specimens of PD effluent will be collected on the day of initiating antibiotic treatment, every 5 days until the day of completing antibiotic treatment, and then 28 days later for the test of LPS level. All patients will be followed for one year after completion of antibiotic therapy for the development of relapsing, recurrent, or repeat peritonitis episodes. Our study would explore the use of detecting LPS in PD effluent as a non-invasive tests for the prediction of relapsing peritonitis.

ELIGIBILITY:
Inclusion Criteria:

at least two of the followings:

1. abdominal pain or cloudy PD effluent;
2. leukocytosis in PD effluent (WBC > 100/ml); and
3. positive Gram-stain or culture from PD effluent

Exclusion Criteria:

* mycobacterial peritonitis
* obvious surgical problems and require laparotomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
relapsing peritonitis | 1 month
  Relapsing peritonitis will be defined as an episode that occurs within 4 weeks of completion of therapy of a prior episode with the same organism (or culture negative in the second episode).
recurrent peritonitis | 1 month
  Recurrent peritonitis will be defined as an episode that occurs within 4 weeks of completion of therapy of a prior episode but with a different organism.
repeat peritonitis | 6 months
  Repeat peritonitis will be defined as an episode that occurs more than 4 weeks after completion of therapy of a prior episode with the same organism.
conversion to long-term hemodialysis | 6 months

SECONDARY OUTCOMES:
peritonitis that requires hospitalization | 6 months
catheter removal | 6 months
death due to peritonitis | 6 months
all cause mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine, Prince of Wales Hospital, Shatin, Hong Kong